CLINICAL TRIAL: NCT03788863
Title: Risk Association of Orofacial Cleft and Glucocorticoids Exposure During Pregnancy: a Meta-analysis
Brief Title: A Study to Learn More About the Relationship Between the Development of a Gap in the Upper Lip (Cleft Lip) or in the Roof of the Mouth (Cleft Palate) in Newborns and the Use of Glucocorticoids by the Mother During Pregnancy: a Meta-analysis
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20638
Record Dates: First submitted 2018-12-13; First posted 2018-12-28 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2019-11

CONDITIONS: Relationship Between the Exposure of Glucocorticoids During Pregnancy and Orofacial Cleft Development
MeSH Terms: interventions — diflucortolone valerate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women exposed to glucocorticoids: Pregnant women exposed to any glucocorticoid or corticosteroid or steroids in early pregnancy or first trimester of pregnancy
  Interventions: Drug: Diflucortolone valerate (BAY866146)
- Non-exposed pregnant women: Women not using any glucocorticoid or corticosteroid or steroids during pregnancy

INTERVENTIONS:
Drug: Diflucortolone valerate (BAY866146) — Follow clinical administration
  Groups: Pregnant women exposed to glucocorticoids

SUMMARY:
Glucocorticoids are drugs that have many effects on body metabolism, raise sugar level in the blood, and reduce inflammation. By applying a statistical technique for combining the findings from a systematic literature review (meta analysis), researchers want to learn more about the relationship of the risk to develop a separation in the roof of the mouth (cleft palate) in newborns and contact with glucocorticoids during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Population: Pregnant women
* Intervention: Any glucocorticoid or corticosteroid or steroids use irrespective of mode of administration
* Comparator: Any/none
* Outcomes: Incidence/ risk of cleft lip/palate in infants
* Study Design:

  * Meta-analysis and systematic literature reviews
  * Observational studies (such as cohort study, case-control study, registries data)
  * Clinical trials - Phase IIb, III, and IV
  * Conference abstracts/posters
* Time period: No time period restriction
* Geography: No geography restriction

Exclusion Criteria:

* Population: Nonpregnant women
* Intervention: Drugs other than glucocorticoid or corticosteroid or steroid
* Outcomes: Incidence/ risk of cleft lip/palate in infants
* Study Design:

  * Animal Study
  * In vitro studies
  * Editorial, letters, comment
  * Clinical trials - Phase I or preclinical
  * Case reports, case series
  * Reviews
* Studies focusing on:

  * Diagnosis and surgical procedure for cleft repair
  * Impact of Increased internal corticosteroids due to stress
  * The relationship between genetic mutations and cleft patients
  * Adverse events for other drugs
  * Safety profiles of glucocorticoid or corticosteroid

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women exposed to any glucocorticoid or corticosteroid or steroids in early pregnancy or first trimester of pregnancy irrespective of mode of administration identified through a systematic review of articles published up to 25 June 2018 by pre-specified inclusion and exclusion criteria. In total 18 observational studies have been selected for this meta-analysis with sample size for individual studies ranging from 106 to 832,636 patients.
Sampling Method: Non-Probability Sample
Enrollment: 99999 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
Incidence of any type of orofacial cleft | Retrospective analysis from 1-Jan-1997 to 25-Jun-2018
  Meta-analysis will be conducted with 18 observational studies. Oral clefts are defined as diagnosis of cleft lip with or without cleft palate or isolated cleft palate.

SECONDARY OUTCOMES:
Potency (mild, moderate, potent, very potent) of glucocorticosteroids | Retrospective analysis from 1-Jan-1997 to 25-Jun-2018
  Potency of glucocorticoid
  * Mild
  * Moderate
  * Potent
  * Very potent
Route of administration of glucocorticosteroids | Retrospective analysis from 1-Jan-1997 to 25-Jun-2018
  Route of administration:
  * Topical
  * Systemic
  * Any other form of use
Types of orofacial cleft | Retrospective analysis from 1-Jan-1997 to 25-Jun-2018
  Types of orofacial cleft
  * Cleft lip (CP)
  * Cleft lip with or without palate (CLP)
  * Cleft palate (CP)
  * Orofacial cleft (OC)

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Germany